CLINICAL TRIAL: NCT02680678
Title: Prevention of Postspinal Hypotension After Spinal Anesthesia for Caesarian Section, the Comparison of Crystalloid and Colloid Infusions and Their Timing Via Perfusion Index and Plethysmographic Variability Index
Brief Title: The Effect of the Timing of Colloid and Crystalloid Infusions on Postspinal Hypotension After Spinal Anesthesia for Caesarian Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, hafize fisun demir, Assistant Professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BAU
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Complications; Anesthesia, Spinal and Epidural, in Pregnancy
MeSH Terms: interventions — succinylated gelatin; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: 4 group of patients were sheduled to receive either kristalloid or kolloid two gropus before and two groups during anesthesia induction
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the outcome accessor and care provider will be aware in which gropu the patient was
Oversight: Data Monitoring Committee: No

ARMS (4):
- Colloid preload (Active Comparator): 20 patients each patient receives 7 ml/kg of gelatin solution (gelofusin) 15 minutes before spinal anesthesia.
  Interventions: Other: Colloid Preload
- Colloid Co-load (Active Comparator): 20 patients each patient receives 7 ml/kg of gelatin solution (gelofusin) beginning with spinal anesthesia.
  Interventions: Other: colloid co-load
- Crystalloid Preload (Active Comparator): 20 patients each patient receives 20 ml/kg of Ringer's lactate solution 15 minutes before spinal anesthesia.
  Interventions: Other: Crystalloid preload
- Crystalloid Co-load (Active Comparator): 20 patients each patient receives 20 ml/kg of Ringer's lactate solution beginning with spinal anesthesia.
  Interventions: Other: Crystalloid Co-load

INTERVENTIONS:
Other: Colloid Preload — preload infusion
  Other Names: Gelofusin
  Arms: Colloid preload
Other: colloid co-load — co-load infusion
  Other Names: gelofusin
  Arms: Colloid Co-load
Other: Crystalloid preload — preload infusion
  Other Names: Ringers lactate solution
  Arms: Crystalloid Preload
Other: Crystalloid Co-load — co-load infusion
  Other Names: Ringers lactate solution
  Arms: Crystalloid Co-load

SUMMARY:
Prevention of postspinal hypotension after spinal anesthesia for caesarian section by use of preoperative or intraoperative volume replacement. The comparison of crystalloid and colloid infusions and their timing via perfusion index and plethysmographic variability index.

DETAILED DESCRIPTION:
To Prevent hypotension fluid replacement is usually used in pregnant patients scheduled for C/S. Different types of fluids can be used in order to achieve this. Also the timing of fluid replacement is important. In the present study patients were separated into 4 groups. Each receiving a one of two fluids in different times. ( Colloid pre-load, colloid co-load, crystalloid co-load and crystalloid pre-load.) The effect of overall hemodynamics and the incidence of hypotension are evaluated. Also peripheric monitors like perfusion index and plethysmographic variability index are evaluated for correlation.

ELIGIBILITY:
Inclusion Criteria:

* pregnant 37-41 weeks
* one fetus
* scheduled for C/S under spinal anesthesia
* accepting to participate

Exclusion Criteria:

* Emergency surgery
* placenta previa
* preeclampsia
* cardiovascular and cerebrovascular comorbidities
* morbid obesity (BMI>40)
* pregnancy weeks <36 and > 41
* The use of vasoconstrictors
* Severe Anemia ( Hb <9 g/dl)
* Refusal or known contraindication for spinal anesthesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of participants in each group who develop hypotension, and correlation between hypotension and Perfusion Index (PI) and Plethysmographic Variability Index (PVI) scores | Measurements will be performed at 5 minute intervals beginning 15 minutes prior to the operation, throughout the whole operation untill the end.
  Hypotension is going tobe measured in mmHG in 5 minute intervals and PI and PVI measurements are also recorded at the same time intervals. A decrease in blood presssure exceeding % 20 of the preoperative basal blood pressure measurement will be recorded as hypotension. The number of patients who develop hypotension will be recorded. Statistic difference will be avaluated between groups. Hypotensive episodes are going to be comparised with the PI and PVI measurements at the same time period and evaluation for correlation will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Hafize Fisun Demir, Principal Investigator — Balikesir University School of Medicine Department of Anesthesia and Reanimation
Locations (1):
- Balikesir University Faculty of Medicine, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No